CLINICAL TRIAL: NCT03412149
Title: Malabsorption and Gut Microbiota Profile Changes After Laparoscopic Mini-Gastric Bypass (MGB) vs Roux-en-Y Gastric Bypass (RYGB): a Prospective Multicenter Comparative Study
Brief Title: Three M Study (Malabsorption, Microbiota, Mini-Gastric Bypass)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianfranco Silecchia, MD PhD Prof. G. Silecchia, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RG11715C7CE1AD8A
Record Dates: First submitted 2017-12-24; First posted 2018-01-26 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Obesity (Disorder)
Keywords: Malabsorption, Mini Gastric Bypass, Roux en Y Gastric Bypass
MeSH Terms: conditions — Obesity; Malabsorption Syndromes | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini Gastric Bypass (Active Comparator): Mini Gastric Bypass: The gastric pouch will be performed starting below the incisura angularis (transverse resection 4 cm) on the lesser curvature (18).Then the stomach will be transected against a 36 Fr bougie up to the gastro-esophageal junction Then 1/3 of the small bowel will be excluded (approximately 200cms) and 3.5-4 cm gastro-jejunostomy will be performed by linear stapler.
  Interventions: Procedure: Mini Gastric Bypass
- Roux en Y Gastric Bypass (Active Comparator): Roux en Y Gastric Bypass: The steps of the standard double loop RYGB technique will be followed (17). The gastric pouch will be created 7 cm from the gastro-esophageal junction to obtain a volume of 30-40 ml, and the length of the alimentary limb will be 150 cm and 3.5-4 cm gastro-jejunostomy will be performed by linear stapler. The length of the biliopancreatic limb will be from 65 to 75 cm beyond the ligament of Treitz. The lengths of both limbs should carefully measured with a graduated instrument. The mesenteric defects will be closed.
  Interventions: Procedure: Roux en Y Gastric Bypass

INTERVENTIONS:
Procedure: Mini Gastric Bypass — Standardization of the techniques will be guaranteed:
  1. Mini Gastric Bypass Arm
  2. Roux en Y Gastric Bypass arm All patients will have intraoperative measurement of the whole length of bowel from Treitz ligament to the ileocecal junction (expected range 6-8 m).The common limb will be therefore about 2/3 of total small bowel length.
  Arms: Mini Gastric Bypass
Procedure: Roux en Y Gastric Bypass — Standardization of the techniques will be guaranteed:
  1. Mini Gastric Bypass Arm
  2. Roux en Y Gastric Bypass arm All patients will have intraoperative measurement of the whole length of bowel from Treitz ligament to the ileocecal junction (expected range 6-8 m).The common limb will be therefore about 2/3 of total small bowel length.
  Arms: Roux en Y Gastric Bypass

SUMMARY:
Bariatric surgery represents the best therapeutic option to induce sustainable weight loss and to solve serious comorbidities improving the life-expectancy and the quality of life. Actually the choice of the procedure is based on the surgeon's and patients preference . Mini gastric bypass(MGB) is an emerging procedure offering excellent results in terms of weight loss and comorbidities (mainly metabolic) control. On the other hand, recent data indicated that the gut microbiota may mediate some of the beneficial effects of bariatric surgery and changes in the composition and diversity of the gut microbiota have been observed after RY Gastric Bypass (RYGB) in humans as well as in mice. However, there are no prospective investigations on Gut Microbiota changes after MGB, despite the procedure is described as "malabsorptive" and there are no studies comparing gut microbiota shift and malabsorption entity in humans after RYGB vs MGB. Thereafter prospective data on the incidence of bile reflux esophageal lesions after MGB are lacking.

The aim of the present multicentric prospective comparative study is to evaluate malabsorption and gut microbiota shift after laparoscopic RYGB vs MGB at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* BMI 40-55 kg/m2
* Non smokers
* Primary Mini Gastric Bypass or Roux en Y Gastric Bypass without any concomitant surgeries except hiatal hernia repair
* Enrollment in the two study groups will be on the basis of patient choice.

Exclusion Criteria:

* Smokers
* Different bowel measurement (plus or minus 10%).
* Conversion to open surgery, reoperation
* Helicobacter Pylori positive previous or current
* Free PPI 4 weeks before 6th month (after surgery)
* Corticosteroids, vitamine E, fish oil treatment 2 months before surgery
* Anti or pre- biotics treatment 2 months before surgery
* Chronic gastrointestinal diseases or syndromes
* Previous bariatric surgery (intragastric balloon excluded)
* Previous resective bowel surgery
* Previous pancreatic surgery
* Previous Hepato BilioPancreatic surgery
* Gallbladder gallstones

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Gut Microbiota | 0-6-12 Months
  To evaluate and compare Roux en Y Gastric Bypass vs Mini Gastric Bypass microbiota profile shift 1 year after surgery and its impact on metabolic and nutritional status after surgery.

SECONDARY OUTCOMES:
Glucagon - like peptide 1 (GLP-1) | 0-12 Months
  To measure GLP-1 plasma level before and 12 months after surgery in MGB vs RYGB patients

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Silecchia, MD PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- ICOT Hospital, Latina, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Milone M, De Placido G, Musella M, Sosa Fernandez LM, Sosa Fernandez LV, Campana G, Di Minno MN, Milone F. Incidence of Successful Pregnancy After Weight Loss Interventions in Infertile Women: a Systematic Review and Meta-Analysis of the Literature. Obes Surg. 2016 Feb;26(2):443-51. doi: 10.1007/s11695-015-1998-7. PMID 26661108
- [Background] Musella M, Apers J, Rheinwalt K, Ribeiro R, Manno E, Greco F, Cierny M, Milone M, Di Stefano C, Guler S, Van Lessen IM, Guerra A, Maglio MN, Bonfanti R, Novotna R, Coretti G, Piazza L. Efficacy of Bariatric Surgery in Type 2 Diabetes Mellitus Remission: the Role of Mini Gastric Bypass/One Anastomosis Gastric Bypass and Sleeve Gastrectomy at 1 Year of Follow-up. A European survey. Obes Surg. 2016 May;26(5):933-40. doi: 10.1007/s11695-015-1865-6. PMID 26341086
- [Background] Campanile FC, Boru CE, Rizzello M, Puzziello A, Copaescu C, Cavallaro G, Silecchia G. Acute complications after laparoscopic bariatric procedures: update for the general surgeon. Langenbecks Arch Surg. 2013 Jun;398(5):669-86. doi: 10.1007/s00423-013-1077-2. Epub 2013 Mar 22. PMID 23519905
- [Background] Rutledge R. The mini-gastric bypass: experience with the first 1,274 cases. Obes Surg. 2001 Jun;11(3):276-80. doi: 10.1381/096089201321336584. PMID 11433900
- [Background] Rutledge R, Walsh TR. Continued excellent results with the mini-gastric bypass: six-year study in 2,410 patients. Obes Surg. 2005 Oct;15(9):1304-8. doi: 10.1381/096089205774512663. PMID 16259892
- [Background] Alexandrou A, Davis PA, Law S, Whooley BP, Murthy SC, Wong J. Esophageal cancer in patients with a history of distal gastrectomy. Arch Surg. 2002 Nov;137(11):1238-42. doi: 10.1001/archsurg.137.11.1238. PMID 12413309
- [Background] Lee WJ, Ser KH, Lee YC, Tsou JJ, Chen SC, Chen JC. Laparoscopic Roux-en-Y vs. mini-gastric bypass for the treatment of morbid obesity: a 10-year experience. Obes Surg. 2012 Dec;22(12):1827-34. doi: 10.1007/s11695-012-0726-9. PMID 23011462
- [Background] Bruzzi M, Rau C, Voron T, Guenzi M, Berger A, Chevallier JM. Single anastomosis or mini-gastric bypass: long-term results and quality of life after a 5-year follow-up. Surg Obes Relat Dis. 2015 Mar-Apr;11(2):321-6. doi: 10.1016/j.soard.2014.09.004. Epub 2014 Sep 16. PMID 25614356
- [Background] Noun R, Skaff J, Riachi E, Daher R, Antoun NA, Nasr M. One thousand consecutive mini-gastric bypass: short- and long-term outcome. Obes Surg. 2012 May;22(5):697-703. doi: 10.1007/s11695-012-0618-z. PMID 22411569
- [Background] Lee WJ, Lee YC, Ser KH, Chen SC, Chen JC, Su YH. Revisional surgery for laparoscopic minigastric bypass. Surg Obes Relat Dis. 2011 Jul-Aug;7(4):486-91. doi: 10.1016/j.soard.2010.10.012. Epub 2010 Oct 30. PMID 21159561
- [Background] Wang W, Wei PL, Lee YC, Huang MT, Chiu CC, Lee WJ. Short-term results of laparoscopic mini-gastric bypass. Obes Surg. 2005 May;15(5):648-54. doi: 10.1381/0960892053923752. PMID 15946455
- [Background] Cavin JB, Voitellier E, Cluzeaud F, Kapel N, Marmuse JP, Chevallier JM, Msika S, Bado A, Le Gall M. Malabsorption and intestinal adaptation after one anastomosis gastric bypass compared with Roux-en-Y gastric bypass in rats. Am J Physiol Gastrointest Liver Physiol. 2016 Sep 1;311(3):G492-500. doi: 10.1152/ajpgi.00197.2016. Epub 2016 Jul 14. PMID 27418681
- [Background] Graessler J, Qin Y, Zhong H, Zhang J, Licinio J, Wong ML, Xu A, Chavakis T, Bornstein AB, Ehrhart-Bornstein M, Lamounier-Zepter V, Lohmann T, Wolf T, Bornstein SR. Metagenomic sequencing of the human gut microbiome before and after bariatric surgery in obese patients with type 2 diabetes: correlation with inflammatory and metabolic parameters. Pharmacogenomics J. 2013 Dec;13(6):514-22. doi: 10.1038/tpj.2012.43. Epub 2012 Oct 2. PMID 23032991
- [Background] Tremaroli V, Karlsson F, Werling M, Stahlman M, Kovatcheva-Datchary P, Olbers T, Fandriks L, le Roux CW, Nielsen J, Backhed F. Roux-en-Y Gastric Bypass and Vertical Banded Gastroplasty Induce Long-Term Changes on the Human Gut Microbiome Contributing to Fat Mass Regulation. Cell Metab. 2015 Aug 4;22(2):228-38. doi: 10.1016/j.cmet.2015.07.009. PMID 26244932
- [Background] Liou AP, Paziuk M, Luevano JM Jr, Machineni S, Turnbaugh PJ, Kaplan LM. Conserved shifts in the gut microbiota due to gastric bypass reduce host weight and adiposity. Sci Transl Med. 2013 Mar 27;5(178):178ra41. doi: 10.1126/scitranslmed.3005687. PMID 23536013
- [Background] Peterson LA, Zeng X, Caufield-Noll CP, Schweitzer MA, Magnuson TH, Steele KE. Vitamin D status and supplementation before and after bariatric surgery: a comprehensive literature review. Surg Obes Relat Dis. 2016 Mar-Apr;12(3):693-702. doi: 10.1016/j.soard.2016.01.001. Epub 2016 Jan 6. PMID 27036669
- [Background] Madan AK, Harper JL, Tichansky DS. Techniques of laparoscopic gastric bypass: on-line survey of American Society for Bariatric Surgery practicing surgeons. Surg Obes Relat Dis. 2008 Mar-Apr;4(2):166-72; discussion 172-3. doi: 10.1016/j.soard.2007.08.006. Epub 2007 Dec 19. PMID 18069071
- [Background] Musella M, Milone M, Deitel M, Kular KS, Rutledge R. What a Mini/One Anastomosis Gastric Bypass (MGB/OAGB) Is. Obes Surg. 2016 Jun;26(6):1322-3. doi: 10.1007/s11695-016-2168-2. No abstract available. PMID 27091050
- [Background] Donini LM, Brunani A, Sirtori A, Savina C, Tempera S, Cuzzolaro M, Spera G, Cimolin V, Precilios H, Raggi A, Capodaglio P; SIO-ISDCA Task Force. Assessing disability in morbidly obese individuals: the Italian Society of Obesity test for obesity-related disabilities. Disabil Rehabil. 2011;33(25-26):2509-18. doi: 10.3109/09638288.2011.575529. Epub 2011 May 4. PMID 21542694

DOCUMENTS (1):
  • Study Protocol (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT03412149/Prot_000.pdf